CLINICAL TRIAL: NCT03603002
Title: Studying the Pathologic and Immunologic Response After Ablative Radiation in Stage I Non-Small Cell Lung Cancer
Brief Title: Pathologic and Immunologic Response After Ablative Radiation in Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J1826; IRB00163415 (Other: JHM IRB)
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer Stage I
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Compare pre- and post-SABR core biopsies of stage I NSCLC tumors to identify SABR-induced immune-mediated tumor recognition based on a significant and specific expansion of T-cell clones using a novel T-cell receptor (TCR) sequencing assay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Stage I NSCLC with SABR Therapy (Experimental): Participants receive stereotactic ablative radiotherapy (SABR) and pre-SABR biopsy as part of standard of care and then receive a post-SABR biopsy after receiving SABR.
  Interventions: Diagnostic Test: Post-SABR Biopsy

INTERVENTIONS:
Diagnostic Test: Post-SABR Biopsy — Post-SABR Biopsy

SUMMARY:
This is a pilot study to compare pre- and post-SABR core biopsies of stage I NSCLC tumors to identify SABR-induced immune-mediated tumor recognition based on a significant and specific expansion of T-cell clones using a novel T-cell receptor (TCR) sequencing assay. This will be coupled with (1) novel genomic analysis of candidate tumor antigens that may be released from the pre-SABR tumor and (2) functional validation assays to screen post-treatment peripheral blood T-cells for reactivity to these released candidate tumor antigens. In addition, cell-based analysis will be used to identify changes in key T-cell infiltrates into the post-SABR tumor.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in the United States. While stereotactic ablative radiotherapy (SABR) is delivered as standard treatment in patients with medically inoperable stage I non-small cell lung cancer (NSCLC), an alarming 30-40% of these patients still develop disease recurrence just outside of the radiation field and deadly distant metastases in their lifetime. Furthermore, since the abscopal response was reported in advanced NSCLC where a systemic cancer response was induced in areas away from the irradiated site when radiation was combined with immunotherapy, multiple clinical trials are currently investigating the role of combining these two modalities. Significantly, how SABR alone increases immunogenicity of a tumor is unknown. There is a critical need to elucidate the mechanism by which SABR alone incites the immune system to better develop future rational combinations of immunotherapy with SABR.

SABR induced cell death will ultimately activate downstream cytotoxic T-cells and cause T-cell influx into the tumor to enhance immunogenic tumor cell kill. This is accomplished with SABR-induced tumor antigen-both mutation-associated neoantigen and tumor-associated antigen- release, priming of downstream cytotoxic T-cells, leading to specific T-cell clonal expansion, and resultant influx of these activated cytotoxic T-cells into the tumor and blood to enhance immune-mediated tumor cell kill.

Herein the investigator proposes a pilot study to compare pre- and post-SABR core biopsies of stage I NSCLC tumors to identify SABR-induced immune-mediated tumor recognition based on a significant and specific expansion of T-cell clones using a novel T-cell receptor (TCR) sequencing assay. This will be coupled with (1) novel genomic analysis of candidate tumor antigens that may be released from the pre-SABR tumor and (2) functional validation assays to screen post-treatment peripheral blood T-cells for reactivity to these released candidate tumor antigens. In addition, cell-based analysis will be used to identify changes in key T-cell infiltrates into the post-SABR tumor.

The results of this pilot study may have the potential to translate into improved systemic outcomes for patients with NSCLC through future integrated trials of immune checkpoint blockade antibodies that specifically relieve the immunosuppression on the T-cell population found to be activated by SABR. Clarifying SABR-induced immune changes in the tumor and blood will identify pathways that may be exploited to enhance systemic immunity to kill micro-metastatic disease and mitigate relapse in the next generation of clinical trials.

Additional corollary imaging studies using dual-energy (DE) computed tomography (CT), a novel imaging modality that improves the material decomposition ability of CTs, may identify new imaging markers for post-SABR treatment response by comparing DE-CT imaging characteristics with SABR fields and pathologic response.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* Age > 18 year
* Confirmed non-small cell lung cancer after initial biopsies
* Patient with accessible tumor for biopsy
* Patient is to have sufficient initial core biopsy samples for tissue analyses
* Stage I lung cancer
* Adequate normal organ and marrow function
* Patient with tumor amenable to SABR treatment as determined by a radiation oncologist
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal subjects. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.

Exclusion Criteria:

* Primary tumors not amenable to serial core biopsies.
* Prior thoracic radiation in the region that will be treated by SABR.
* Patient may not be receiving any other concurrent investigational agents or chemotherapy.
* Patient may not be receiving or received immunotherapy.
* Patients may not be on or use steroids within 14 days before radiation, and from the duration of radiation to the time of the post-SABR biopsies and blood samples.
* Female patients who are pregnant from screening to completion of SABR

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2025-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khinh Ranh Voong, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stage I NSCLC With SABR Therapy
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stage I NSCLC With SABR Therapy
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: Years] | 75 [66 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Examine the T-cell Receptor Profile Changes Induced in the Tumor After SABR
Description: T-cell receptor (TCR) profile changes in the tumor using TCR sequencing.
Time Frame: Baseline to up to 7 days after SABR treatment
Population: None of the core-needle samples were able to be analyzed and no data was collected from samples.
Arm/Group | Stage I NSCLC With SABR Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Evaluate Candidate Tumor Antigens Released From the Tumor by SABR
Description: Candidate tumor antigens, mutation associated neo-antigens (MANAs), and tumor associated neo-antigens, (TAAs) released from the tumor by SABR
Time Frame: post-SABR
Population: None of the core-needle samples were able to be analyzed and no data was collected from samples.
Arm/Group | Stage I NSCLC With SABR Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Semiquantitative Scoring System to Describe the Influx of Key Tumor Infiltrating Lymphocytes in the Tumor After SABR.
Description: Semiquantitative immunohistochemistry scoring system was used to evaluate pathological changes, immune-cell populations (CD8, FoxP3), within the tumor. Semiquantitative scoring system: 0 None, 1: 1-5, 2: 6-10, 3: 11-20, 4: 21 or more positive cells per high powered field (400x). Score for each participant is reported.
Time Frame: 5 to 7 day post SABR
Population: Scores for each participant is reported.
Measure: Number; unit: score on a scale
Arm/Group | Stage I NSCLC With SABR Therapy
Number analyzed (Participants) | 6
score on a scale
  Participant 1, CD8: number analyzed (Participants) | 1
  Participant 1, CD8 | 0
  Participant 2, CD8: number analyzed (Participants) | 1
  Participant 2, CD8 | 0
  Participant 3, CD8: number analyzed (Participants) | 1
  Participant 3, CD8 | 0
  Participant 4, CD8: number analyzed (Participants) | 1
  Participant 4, CD8 | NA — No tumor or minimal detected on slide
  Participant 5, CD8: number analyzed (Participants) | 1
  Participant 5, CD8 | NA — No tumor or minimal detected on slide
  Participant 6, CD8: number analyzed (Participants) | 1
  Participant 6, CD8 | 1
  Participant 1, FoxP3: number analyzed (Participants) | 1
  Participant 1, FoxP3 | 0
  Participant 2, FoxP3: number analyzed (Participants) | 1
  Participant 2, FoxP3 | NA — No tumor or minimal detected on slide
  Participant 3, FoxP3: number analyzed (Participants) | 1
  Participant 3, FoxP3 | 0
  Participant 4, FoxP3: number analyzed (Participants) | 1
  Participant 4, FoxP3 | NA — No tumor or minimal detected on slide
  Participant 5, FoxP3: number analyzed (Participants) | 1
  Participant 5, FoxP3 | NA — No tumor or minimal detected on slide
  Participant 6, FoxP3: number analyzed (Participants) | 1
  Participant 6, FoxP3 | 1

4. Secondary Outcome: Detection of Peripheral Neoantigen-specific T-cell Responses and Dynamics After SABR.
Description: Assessed by the Mutation-Associated Neoantigen Functional Expansion of Specific T-cells (MANAFEST) assay. Number of participants where a peripheral neoantigen-specific T-cell responses and dynamics was detected is reported.
Time Frame: Within one year after SABR
Population: Four patients had sufficient paired pre- and post-SABR tumor and blood samples for analysis to identify antigen-specific TCRs in the blood.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage I NSCLC With SABR Therapy
Number analyzed (Participants) | 4
Participants | 2

5. Secondary Outcome: Dual-energy (DE) CT Imaging Characteristics After SABR
Description: Dual-energy (DE) CT imaging characteristics after SABR. Evaluate relationship between dual-energy (DE) CT imaging characteristics, radiation dose, and early post-SABR pathologic outcomes after treatment with SABR.
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2026-03

6. Secondary Outcome: Number of Participants With Grade 2+ Toxicity Events
Description: Patients with grade 2+ toxicity measured by NCIs Common Terminology Criteria for Adverse Events (CTCAE 4.0), due to post-SABR biopsy.
Time Frame: Pre-SABR, Post-SABR, 3, 6, 9 and 12 months.
Measure: Number; unit: Participants
Arm/Group | Stage I NSCLC With SABR Therapy
Number analyzed (Participants) | 6
Participants | 0

7. Secondary Outcome: Semiquantitative Scoring System to Describe the Influx of Key Tumor Infiltrating Lymphocytes Within the Peritumoral Stoma After SABR.
Description: Semiquantitative immunohistochemistry scoring system was used to evaluate pathological changes, (CD8, FoxP3, PD-L1/PD-1) expression within the peritumoral stoma after SABR. Semiquantitative scoring system: 0 None, 1: 1-5, 2: 6-10, 3: 11-20, 4: 21 or more positive cells per high powered field (400x). Score for each participant is reported.
Time Frame: 5 to 7 day post SABR
Population: Scores for each participant is reported
Measure: Number; unit: score on a scale
Arm/Group | Stage I NSCLC With SABR Therapy
Number analyzed (Participants) | 6
score on a scale
  Participant 1, CD8: number analyzed (Participants) | 1
  Participant 1, CD8 | 4
  Participant 2, CD8: number analyzed (Participants) | 1
  Participant 2, CD8 | 2
  Participant 3, CD8: number analyzed (Participants) | 1
  Participant 3, CD8 | 3
  Participant 4, CD8: number analyzed (Participants) | 1
  Participant 4, CD8 | 4
  Participant 5, CD8: number analyzed (Participants) | 1
  Participant 5, CD8 | NA — No tumor or minimal detected on slide
  Participant 6, CD8: number analyzed (Participants) | 1
  Participant 6, CD8 | 3
  Participant 1, FoxP3: number analyzed (Participants) | 1
  Participant 1, FoxP3 | 3
  Participant 2, FoxP3: number analyzed (Participants) | 1
  Participant 2, FoxP3 | 3
  Participant 3, FoxP3: number analyzed (Participants) | 1
  Participant 3, FoxP3 | 1
  Participant 4, FoxP3: number analyzed (Participants) | 1
  Participant 4, FoxP3 | 3
  Participant 5, FoxP3: number analyzed (Participants) | 1
  Participant 5, FoxP3 | NA — No tumor or minimal detected on slide
  Participant 6, FoxP3: number analyzed (Participants) | 1
  Participant 6, FoxP3 | 3
  Participant 1, PD1: number analyzed (Participants) | 1
  Participant 1, PD1 | 3
  Participant 2, PD1: number analyzed (Participants) | 1
  Participant 2, PD1 | 2
  Participant 3, PD1: number analyzed (Participants) | 1
  Participant 3, PD1 | 2
  Participant 4, PD1: number analyzed (Participants) | 1
  Participant 4, PD1 | 4
  Participant 5, PD1: number analyzed (Participants) | 1
  Participant 5, PD1 | NA — No tumor or minimal detected on slide
  Participant 6, PD1: number analyzed (Participants) | 1
  Participant 6, PD1 | 3

ADVERSE EVENTS:
Time Frame: Pre-SABR, Post-SABR, 3, 6, 9 and 12 months.
Arm/Group | Stage I NSCLC With SABR Therapy
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage I NSCLC With SABR Therapy (N=6)
Anemia (Psychiatric disorders) | 1 (1)
Anorexia (Psychiatric disorders) | 2 (3)
anxiety (Psychiatric disorders) | 4 (5)
Bronchial Infection (Infections and infestations) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (General disorders) | 6 (14)
Difficulty swallowing (General disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (13)
Fatigue (General disorders) | 6 (10)
Headache (General disorders) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Peripheral Sensory Neuropathy (Nervous system disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT03603002/Prot_SAP_000.pdf